CLINICAL TRIAL: NCT07400835
Title: The ENDOMETRIAL Study: EvaluatioN of DNA methylatiOn Markers for EndomeTrial Cancer Risk-stratification Using Patient-collected urIne and vAginal Samples and Clinician-collected Cervical Samples From Women With Postmenopausal bLeeding
Brief Title: Evaluation of DNA Methylation Markers for Endometrial Cancer Risk-stratification Using Patient-collected Urine and Vaginal Samples and Clinician-collected Cervical Samples From Women With Postmenopausal Bleeding
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other); University of Southern Denmark (Other); University Clinic for Cancer Screening, Department of Public Health Programmes, Randers Regional Hospital, Central Denmark Region (Unknown); Region of Southern Denmark (Other); Amsterdam UMC (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: endometrial-PMB-stúdy
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postmenopausal Bleeding
Keywords: DNA methylation; Postmenopausal bleeding; Endometrial Cancer; Patient-collected urine samples; patient-collected vaginal samples; cervical samples
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Patient-collected urine and vaginal samples, and clinician-collecteed cervical samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with postmenopausal bleeding: Women referred for diagnostic evaluation to gynaecological departments for endometrial cancer due to postmenopausal bleeding
  Interventions: Diagnostic Test: DNA-methylation testing in patient-collected urine and vaginal samples and clinician-collected cervical samples

INTERVENTIONS:
Diagnostic Test: DNA-methylation testing in patient-collected urine and vaginal samples and clinician-collected cervical samples — DNA-methylation testing of methylation markers CDO1, GHSR and ZIC1 for patient-collected vaginal samples, GHSR, CDH13 and SST for patient-collected urine samples and CDH13 + CDO1 + ZIC1 for clinician-collected cervical samples.

SUMMARY:
The goal of this observational study is to investigate the clinical utility of DNA-methylation testing in urine and vaginal samples collected by patients and cervical samples collected by clinicians, to determine the risk of endometrial cancer in symptomatic women with postmenopausal bleeding. The study aims to answer the following research questions:

* What is the diagnostic accuracy of DNA methylation testing in urine, vaginal and cervical samples compared to traditional TVUS for endometrial cancer detection?
* What is the 2 year risk of EC among women testing negative on TVUS and/or DNA methylation tests or those testing positive on methylation only?

Researchers will compare DNA methylation testing in patient-collected urine and vaginal samples as well as in clinician-collected cervical samples, with the traditional diagnostic pathway for women with PMB, which includes TVUS-evaluation, and when indicated by abnormal TVUS findings, endometrial biopsy according to clinical guidelines.

Participants will

* take a urine and vaginal sample
* Have a cervical sample collected by a clinician
* Undergo TVUS evaluation according to clinical guidelines
* If TVUS shows thickened endometrium (≥ 5 mm) and/or irregularity, an endometrial biopsy will be collected according to clinical guidelines
* Participants will fill out a questionnaire regarding acceptability and preferences of sampling methods and answer a lifestyle questionnaire.

DETAILED DESCRIPTION:
BACKGROUND:

Endometrial cancer (EC) incidence is raising and is the fourth most common cancer type in women worldwide with about 417,000 new cases and 90,000 deaths annually. Moreover, EC is the most common gynaecological cancer in developed countries including Denmark with about 800 new cases and 90 deaths yearly. Early diagnosis is essential since the prognosis for women with an advanced EC stage is poor. No screening exists for EC and the most commonly observed clinical symptom is post-menopausal bleeding (PMB), which is a common condition affecting about 11% of postmenopausal women. Because 90% of EC cases, are preceded by PMB, referral for specialized gynaecological care through cancer patient pathways is indicated for all Danish women with PMB, causing anxiety among women and high health-care costs. However, only 5-10% of women presenting with PMB have EC. Worldwide, transvaginal ultrasound (TVUS) evaluation of the endometrium (cut-off: thickness ≥5mm and/or irregular lining of the uterine cavity) is used to identify women with PMB who have the highest cancer risk and therefore require an endometrial biopsy with or without hysteroscopy. While TVUS evaluation is highly sensitive (94.8%) it suffers from low specificity (51%) causing high numbers of unnecessary invasive procedures in healthy women. Moreover, the diagnostic program depends on skilled specialists for ultrasound evaluation, endometrial sampling as well as histopathological examination. This reinforces the clinical urgent and unmet need for a simpler, non-invasive, user-provided and more specific test to aid EC diagnosis.

This study aims to determine whether DNA methylation testing in patient-collected urine and vaginal samples is a clinically safe non-invasive alternative to determine EC risk. Testing for elevated DNA hypermethylation levels of cancer-specific genes has been demonstrated to provide a promising biomarker for detection of early-stage cancers, including cervical and endometrial cancer. DNA hypermethylation has been linked to silencing of tumour suppressor genes, thereby contributing to cancer development. Biologically, the ability to use vaginal and urine material for EC detection by DNA methylation testing is explained by local shedding of EC-derived DNA and cell fragments into the vaginal debris and urine as well as transrenal excretion of tumour-shedded circulating DNA into the urine.

Mainly small proof-of-concepts and case-controls studies have shown feasibility to detect EC using DNA methylation testing in plasma, self-collected vaginal samples, and clinician-collected cervical scrapes. However, the first paper reporting on the diagnostic value of DNA methylation analysis in vaginal samples and urine as a liquid biopsy for EC was just published by co-supervisor Prof. Steenbergen last year. Here, case-control data revealed excellent diagnostic performance of EC-specific DNA methylation markers in patient-collected urine and vaginal samples with sensitivities of 89-90% and specificities of 90-92% for EC detection using markers panels including: CDH13, GHSR, SST, CDO1, and ZIC1.

Only one prospective cohort study has compared the diagnostic performance of DNA methylation testing in clinician-collected cervicovaginal samples with the conventional TVUS evaluation in terms of detecting the presence or absence of EC in women aged 45+ with abnormal uterine bleeding. The results demonstrated the WID-qEC DNA methylation test (markers: ZSCAN12 and GYPC) to have equal sensitivity (90.9%) and superior specificity (92.1 vs 79.1%) as compared to TVUS evaluation.

However, this will be the first study to compare DNA methylation testing in patient-collected urine and vaginal samples to TVUS evaluation.

STUDY DESIGN: Comparative diagnostic accuracy study, comparing diagnostic test methods at the time of diagnosis as well as the long-term safety after two years.

MATERIALS AND METHODS:

The vaginal, urine and cervical samples will be stored in a biobank at the Dept. of Pathology, Randers Regional Hospital (RHR) until shipment for DNA methylation testing analysis using quantitative methylation-specific PCR (qMSP) in Prof. Steenbergens' laboratory at Amsterdam University Medical Centre, The Netherlands. All samples will be tested for methylation markers, three for vaginal samples (CDO1, GHSR, ZIC1), three for urine (GHSR, CDH13, SST) and three for cervical samples (CDH13 + CDO1 + ZIC1). Results on TVUS evaluation and endometrial biopsies will be retrieved from the nationwide Danish Pathology Databank and the electronic patient journal linked to the patient through the Civil Registration System in Denmark, where all residents have a unique 10-cipher code (CPR-number), to which all health data is linked.

AIMs:

1. To determine the diagnostic accuracy of DNA methylation testing in patient-collected full-void urine and vaginal samples, as well as clinician-collected cervical samples to detect EC among women with postmenopausal bleeding, and 2) to compare the diagnostic test accuracy of DNA methylation to the current diagnostic evaluation with TVUS.
2. To assess the preferences and experiences for type of diagnostic evaluation, including urine, vaginal and cervical samples and TVUS.

HYPOTHESES:

1. DNA methylation testing in urine samples can detect EC with comparable sensitivity and superior specificity as compared to TVUS and with higher accuracy than DNA methylation testing in vaginal and cervical samples.
2. DNA methylation analysis in urine samples will have a long-term negative EC risk after 2 years equivalent to TVUS, but better than vaginal and cervical samples.

RESEARCH PLAN AND FEASIBILITY The study will be conducted in collaboration between University Clinic for Cancer Screening, Dept. of Public Health Programmes, Dept. of Pathology, RHR and with gynaecological departments in Central Denmark (Randers and Aarhus) and Southern Denmark Region (Odense) working as inclusion sites. State-of-the-art laboratory facilities are in place at Prof. Steenbergen's laboratory at Amsterdam UMC, supporting the feasibility of the studies.

PERSPECTIVES AND COMMUNICATION If successful, the research will have international impact and result in a novel diagnostic tool that will differentiate between women with PMB who do or do not need specialist referral through cancer patients' pathways to have invasive endometrial biopsies. This will facilitate timely diagnosis, lower the anxiety among patients, and reducing the pressure on the health-care system. Results will be published in international peer-reviewed journals and presented at conferences and will be concluded with a PhD dissertation. The results will be distributed to relevant clinical fora and implemented in national as well as international guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal bleeding (defined as vaginal bleeding after absence of periods for ≥ 12 months) undergoing diagnostic evaluation for EC at gynaecological departments
* Treated in Central Denmark Region or Southern Denmark Region, Denmark
* Able to provide written consent for participation
* Able to read and understand Danish

Exclusion Criteria:

* Other concurrent cancer diagnosis besides diagnostic evaluation for postmenopausal bleeding
* Withdrawal of consent
* Hysterectomized

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with postmenopausal bleeding undergoing diagnostic evaluation for endometrial cancer will be recruited from Department of Obstetrics and Gynaecology, Aarhus University Hospital, Randers Regional Hospital, Central Denmark Region, and Odense University Hospital, Southern Denmark Region, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2028-02-02 (Estimated); Study Completion 2030-02-02 (Estimated)

PRIMARY OUTCOMES:
Area under the Curve (AUC) | At the time of enrollment and to the time of diagnosis
  The performance of each methylation marker panels in urine, vaginal and cervical samples and the TVUS will be evaluated by area Under the Curve with 95% CIs.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Tranberg, PhD, Principal Investigator — University Clinic for Cancer Screening, Department of Public Health Programmes, Randers Regional Hospital
Locations (3):
- Denmark (3):
  - Department of Obstetrics and Gynaecology, Aarhus University Hospital, Aarhus N
  - Department of Obstetrics and Gynaecology, Odense University Hospital, Odense
  - Department of Obstetrics and Gynaecology, Randers Regional Hospital, Randers

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Crosbie EJ, Kitson SJ, McAlpine JN, Mukhopadhyay A, Powell ME, Singh N. Endometrial cancer. Lancet. 2022 Apr 9;399(10333):1412-1428. doi: 10.1016/S0140-6736(22)00323-3. PMID 35397864
- [Background] Engholm G, Ferlay J, Christensen N, Bray F, Gjerstorff ML, Klint A, Kotlum JE, Olafsdottir E, Pukkala E, Storm HH. NORDCAN--a Nordic tool for cancer information, planning, quality control and research. Acta Oncol. 2010 Jun;49(5):725-36. doi: 10.3109/02841861003782017. PMID 20491528
- [Background] Gustafson LW, Booth BB, Kahlert J, Ortoft G, Mejlgaard E, Clarke MA, Wentzensen N, Rositch AF, Hammer A. Trends in hysterectomy-corrected uterine cancer mortality rates during 2002 to 2015: mortality of nonendometrioid cancer on the rise? Int J Cancer. 2021 Feb 1;148(3):584-592. doi: 10.1002/ijc.33219. Epub 2020 Aug 17. PMID 32683690
- [Background] Long B, Clarke MA, Morillo ADM, Wentzensen N, Bakkum-Gamez JN. Ultrasound detection of endometrial cancer in women with postmenopausal bleeding: Systematic review and meta-analysis. Gynecol Oncol. 2020 Jun;157(3):624-633. doi: 10.1016/j.ygyno.2020.01.032. Epub 2020 Jan 31. PMID 32008795
- [Background] Astrup K, Olivarius Nde F. Frequency of spontaneously occurring postmenopausal bleeding in the general population. Acta Obstet Gynecol Scand. 2004 Feb;83(2):203-7. doi: 10.1111/j.0001-6349.2004.00400.x. PMID 14756741
- [Background] Herzog C, Marin F, Jones A, Evans I, Reisel D, Redl E, Schreiberhuber L, Paytubi S, Pelegrina B, Carmona A, Peremiquel-Trillas P, Frias-Gomez J, Pineda M, Brunet J, Ponce J, Matias-Guiu X, de Sanjose S, Alemany L, Olaitan A, Wong M, Jurkovic D, Crosbie EJ, Rosenthal AN, Bjorge L, Zikan M, Dostalek L, Cibula D, Sundstrom K, Dillner J, Costas L, Widschwendter M. A Simple Cervicovaginal Epigenetic Test for Screening and Rapid Triage of Women With Suspected Endometrial Cancer: Validation in Several Cohort and Case/Control Sets. J Clin Oncol. 2022 Nov 20;40(33):3828-3838. doi: 10.1200/JCO.22.00266. Epub 2022 Aug 24. PMID 36001862
- [Background] Morice P, Leary A, Creutzberg C, Abu-Rustum N, Darai E. Endometrial cancer. Lancet. 2016 Mar 12;387(10023):1094-1108. doi: 10.1016/S0140-6736(15)00130-0. Epub 2015 Sep 6. PMID 26354523
- [Background] van den Helder R, Wever BMM, van Trommel NE, van Splunter AP, Mom CH, Kasius JC, Bleeker MCG, Steenbergen RDM. Non-invasive detection of endometrial cancer by DNA methylation analysis in urine. Clin Epigenetics. 2020 Nov 3;12(1):165. doi: 10.1186/s13148-020-00958-7. PMID 33143739
- [Background] Kulis M, Esteller M. DNA methylation and cancer. Adv Genet. 2010;70:27-56. doi: 10.1016/B978-0-12-380866-0.60002-2. PMID 20920744
- [Background] Hentschel AE, van den Helder R, van Trommel NE, van Splunter AP, van Boerdonk RAA, van Gent MDJM, Nieuwenhuijzen JA, Steenbergen RDM. The Origin of Tumor DNA in Urine of Urogenital Cancer Patients: Local Shedding and Transrenal Excretion. Cancers (Basel). 2021 Jan 31;13(3):535. doi: 10.3390/cancers13030535. PMID 33572525
- [Background] den Helder RV, Wever BM, van Trommel JA, Ket JC, Bleeker MC, Steenbergen RD, van Trommel NE. DNA methylation markers for endometrial cancer detection in minimally invasive samples: a systematic review. Epigenomics. 2020 Sep;12(18):1661-1672. doi: 10.2217/epi-2020-0164. Epub 2020 Sep 17. PMID 32938224
- [Background] Fiegl H, Gattringer C, Widschwendter A, Schneitter A, Ramoni A, Sarlay D, Gaugg I, Goebel G, Muller HM, Mueller-Holzner E, Marth C, Widschwendter M. Methylated DNA collected by tampons--a new tool to detect endometrial cancer. Cancer Epidemiol Biomarkers Prev. 2004 May;13(5):882-8. PMID 15159323
- [Background] Doufekas K, Hadwin R, Kandimalla R, Jones A, Mould T, Crowe S, Olaitan A, Macdonald N, Fiegl H, Wik E, Salvesen HB, Widschwendter M. GALR1 methylation in vaginal swabs is highly accurate in identifying women with endometrial cancer. Int J Gynecol Cancer. 2013 Jul;23(6):1050-5. doi: 10.1097/IGC.0b013e3182959103. PMID 23727823
- [Background] Kim GE, Kweon SS, Lee JS, Lee JH, Nam JH, Choi C. Quantitative assessment of DNA methylation for the detection of cervical and endometrial adenocarcinomas in liquid-based cytology specimens. Anal Quant Cytopathol Histpathol. 2012 Aug;34(4):195-203. PMID 23016466
- [Background] De Strooper LM, van Zummeren M, Steenbergen RD, Bleeker MC, Hesselink AT, Wisman GB, Snijders PJ, Heideman DA, Meijer CJ. CADM1, MAL and miR124-2 methylation analysis in cervical scrapes to detect cervical and endometrial cancer. J Clin Pathol. 2014 Dec;67(12):1067-71. doi: 10.1136/jclinpath-2014-202616. Epub 2014 Oct 3. PMID 25281766
- [Background] Bakkum-Gamez JN, Sherman ME, Slettedahl SW, Mahoney DW, Lemens MA, Laughlin-Tommaso SK, Hopkins MR, VanOosten A, Shridhar V, Staub JK, Cao X, Foote PH, Clarke MA, Burger KN, Berger CK, O'Connell MC, Doering KA, Podratz KC, DeStephano CC, Schoolmeester JK, Kerr SE, Wentzensen N, Taylor WR, Kisiel JB. Detection of endometrial cancer using tampon-based collection and methylated DNA markers. Gynecol Oncol. 2023 Jul;174:11-20. doi: 10.1016/j.ygyno.2023.04.014. Epub 2023 May 2. PMID 37141817
- [Background] Wever BMM, van den Helder R, van Splunter AP, van Gent MDJM, Kasius JC, Trum JW, Verhoeve HR, van Baal WM, Hulbert A, Verhoef L, Heideman DAM, Lissenberg-Witte BI, van Trommel NE, Steenbergen RDM, Bleeker MCG. DNA methylation testing for endometrial cancer detection in urine, cervicovaginal self-samples and cervical scrapes. Int J Cancer. 2023 Jul 15;153(2):341-351. doi: 10.1002/ijc.34504. Epub 2023 Mar 23. PMID 36912267
- [Background] Snoek BC, Splunter APV, Bleeker MCG, Ruiten MCV, Heideman DAM, Rurup WF, Verlaat W, Schotman H, Gent MV, Trommel NEV, Steenbergen RDM. Cervical cancer detection by DNA methylation analysis in urine. Sci Rep. 2019 Feb 28;9(1):3088. doi: 10.1038/s41598-019-39275-2. PMID 30816167
- [Background] Guerrero-Preston R, Valle BL, Jedlicka A, Turaga N, Folawiyo O, Pirini F, Lawson F, Vergura A, Noordhuis M, Dziedzic A, Perez G, Renehan M, Guerrero-Diaz C, De Jesus Rodriguez E, Diaz-Montes T, Rodriguez Orengo J, Mendez K, Romaguera J, Trock BJ, Florea L, Sidransky D. Molecular Triage of Premalignant Lesions in Liquid-Based Cervical Cytology and Circulating Cell-Free DNA from Urine, Using a Panel of Methylated Human Papilloma Virus and Host Genes. Cancer Prev Res (Phila). 2016 Dec;9(12):915-924. doi: 10.1158/1940-6207.CAPR-16-0138. Epub 2016 Sep 26. PMID 27671338
- [Background] Van Keer S, van Splunter AP, Pattyn J, De Smet A, Herzog SA, Van Ostade X, Tjalma WAA, Ieven M, Van Damme P, Steenbergen RDM, Vorsters A. Triage of human papillomavirus infected women by methylation analysis in first-void urine. Sci Rep. 2021 Apr 12;11(1):7862. doi: 10.1038/s41598-021-87329-1. PMID 33846517
- [Background] Evans I, Reisel D, Jones A, Bajrami A, Nijjar S, Solangon SA, Arora R, Redl E, Schreiberhuber L, Ishaq-Parveen I, Rotharmel J, Herzog C, Jurkovic D, Widschwendter M. Performance of the WID-qEC test versus sonography to detect uterine cancers in women with abnormal uterine bleeding (EPI-SURE): a prospective, consecutive observational cohort study in the UK. Lancet Oncol. 2023 Dec;24(12):1375-1386. doi: 10.1016/S1470-2045(23)00466-7. Epub 2023 Nov 6. PMID 37944542
- [Background] Erichsen R, Lash TL, Hamilton-Dutoit SJ, Bjerregaard B, Vyberg M, Pedersen L. Existing data sources for clinical epidemiology: the Danish National Pathology Registry and Data Bank. Clin Epidemiol. 2010 Aug 9;2:51-6. doi: 10.2147/clep.s9908. PMID 20865103